CLINICAL TRIAL: NCT03657277
Title: Characterizing Epidermal Responses Following Micropatch Application at Various Body Sites in Human Subjects
Brief Title: Micropore Closure Kinetics at Various Body Sites
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Nicole K Brogden, Associate Professor, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 201806039
Record Dates: First submitted 2018-08-30; First posted 2018-09-05 (Actual); Results first posted 2021-07-28 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Healthy
Keywords: Peer Reviewed Research

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Micropatch Application (Other): This is the only study arm, which all participants complete. Five sites each on each the upper arm, forearm, and abdomen will be identified. Baseline measurements of trans-epidermal water loss, electrical resistance, hydration, and skin color will be made. Micropatches will be applied at three sites (at each body location). This only occurs on the first study day. Trans-epidermal water loss and electrical resistance are re-measured immediately after micropatch application. The sites will be covered with a small patch secured with medical tape. One site at each location will just be covered with a patch. The last site will not have micropatch application or patches. Electrical resistance will be re-measured at all sites for 3 days. Measurements from the 4th and 5th sites allow each subject to serve as their own control in data analysis.
  Interventions: Device: Micropatch

INTERVENTIONS:
Device: Micropatch — Each micropatch contains 50 tiny projections (800 um in length)

SUMMARY:
The study to be performed will define the rate of skin barrier recovery following micropatch application to the skin on the upper arm, volar forearm, and abdomen in healthy subjects.

DETAILED DESCRIPTION:
Transdermal drug delivery (by way of patches that adhere to the skin and deliver drug in a time-dependent fashion) allows for systemic drug delivery through the skin, while avoiding many of the side effects and challenges associated with oral or intravenous drug delivery. One significant challenge limiting the number of drug compounds that can be transdermally delivered is the hydrophobic nature of the skin, which provides a barrier against absorption of drug molecules. Micropatches are a specialized type of patch that help drug molecules to cross the skin by creating micron-sized channels (also called micropores) in the skin, which makes the skin more permeable. Micropatches have been safely used in hundreds of patients for administration of drugs and vaccines through the skin. Studies have demonstrated that micropatch application is relatively painless and well-tolerated by most patients.

Following micropatch application, the skin must reseal the micropores in order to restore the skin's full barrier function. In young healthy individuals this process takes approximately 48 to 72 hours when the skin is covered by an occlusive patch. The timeframe is longer in older individuals who are >65 years of age. As evidenced by these age-related differences in restoration of skin barrier function, biological variation can have a significant effect on the skin's response after micropatch application. There are almost no data available regarding how race and ethnicity affect skin response to micropatch application. It is crucial to better understand how the rates of restoring barrier function vary in different racial/ethnic populations. This is very important for reducing potential for variability in drug delivery when new micropatches are developed in the future for treating diseases.

In this study researchers are examining skin characteristics and response to micropatch application, but there will be no drugs delivered in this study. Hydration and color will be measured to characterize the epidermal properties of individuals of different self-identified race and ethnicity. Measurements of trans-epidermal water loss and electrical impedance will be used to evaluate the formation of micropores in the skin; the electrical impedance measurements will be used to calculate the rate of barrier function repair. All of these skin characteristics can be measured using noninvasive methods that are quick and painless.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 50 years of age
* Healthy, non-obese men and women
* Identify as African American or Black, Asian, Hispanic or Latino, Caucasian/White, bi-/multiracial or other

Exclusion Criteria:

* Unable to give consent
* Severe general allergies requiring chronic treatment with steroids or antihistamines
* Previous adverse reaction to micropatch application
* Previous history of keloids
* Known allergy or adverse reaction to medical tape/adhesive or aloe vera
* Any inflammatory diseases of the skin; psoriasis, atopic dermatitis, and blistering skin disorders
* Diseases associated with altered immune function (including but not limited to: rheumatoid arthritis, diabetes, lupus, HIV/AIDS)
* Any subjects taking medication that impairs the immune system (including but not limited to corticosteroids, TNF inhibitors, monoclonal antibodies, chemotherapy agents)
* Any current malignancy or history of malignancy present at the micropatch application sites
* Eczema or scaling present at the application sites
* Any current inflammation or irritation present at the application sites (including but not limited to: rash, inflammation, erythema, edema, blisters)
* BMI>29.9
* Uncontrolled mental illness that would, in the opinion of the physician, affect the subject's ability to understand or reliably participate in the study
* Subjects taking medications in the following therapeutic classes will be excluded: HMGCoA reductase inhibitors ("statins"), oral or topical steroids, oral antibiotics, topical antibiotics at the micropatch application sites, topical antihistamines at the micropatch application sites, beta-blockers, and systemic or topical NSAIDS/analgesics/anti-inflammatories. A subject who has recently used oral or topical steroids, antibiotics, antihistamines, or analgesics may be enrolled if sufficient time has passed since the last dose (as determined by a member of the study team).
* Any subjects that are pregnant/nursing will be excluded from participation.
* Any condition that would, in the opinion of the study team, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-03-18 (Actual); Study Completion 2021-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Brogden, PharmD, PhD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment on this study was open from October 2018 to March 2020. Study procedures were conducted at the University of Iowa Hospitals and Clinics in the Clinical Research Clinic by members of the research staff.
Pre-assignment Details: Subjects were screened after consenting to participate in the study. 2 of our 46 participants met exclusionary criteria after consenting. 1 of 46 participants signed the consent and stopped returning communication with study staff and was withdrawn from the study due to lack of follow-up. 8 of 46 were withdrawn from the study, prior to completing any visits, as a result of the closure of our clinical research unit due to the COVID-19 pandemic.
Period: Overall Study
Arm/Group | Micropatch Application
Started | 46
Completed | 35
Not Completed | 11
Not completed — Physician Decision | 2
Not completed — Lost to Follow-up | 1
Not completed — Covid-19 Research Halt at University of Iowa-Withdrawal of subjects | 8

BASELINE CHARACTERISTICS:
Arm/Group | Micropatch Application
Number analyzed (Participants) | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 46
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 25.0 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic/Latino | 7
  Caucasian/White | 12
  Asian | 10
  African American/Black | 11
  Other-Pacific Islander | 1
  Bi-/Multiracial | 5

OUTCOME MEASURES:

1. Primary Outcome: Micropore Re-sealing Kinetics
Description: The time required for the skin barrier to be restored after micropatch application at 3 sites on the body will be determined using electrical resistance measurements. Differences in the skin electrical resistance will be determined through measurements made every day with skin electrodes attached to an impedance meter. These data for micropore re-sealing are only collected from the micropatch sites.
Time Frame: Four Days
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Micropatch Application
Number analyzed (Participants) | 35
hours
  Forearm | 58.29 (16.76)
  Upper arm | 60.34 (14.69)
  Abdomen | 63.09 (13.13)

2. Secondary Outcome: Change in Trans-epidermal Water Loss
Description: Percent change from baseline trans-epidermal water loss will be calculated after micropatch application at each body site, and these data are only collected from the micropatch sites. Percent change is calculated as (trans-epidermal water loss after micropatch application/baseline trans-epidermal water loss) x 100.
Time Frame: Baseline (Day 0) and post micropatch application (Day 0)
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Micropatch Application
Number analyzed (Participants) | 35
percent change
  Forearm | 243.96 (126.33)
  Upper arm | 264.46 (151.20)
  Abdomen | 225.47 (137.67)

3. Secondary Outcome: Skin Color Groups
Description: Lightness/darkness of the skin is measured with a tristimulus colorimeter and reported in a unitless value called L*. Higher L* values denote lighter skin, while lower L* values denote darker skin. Data are calculated as the mean of measurements from all sites on the abdomen, and subjects are grouped into categories based on ranges of L*.
Time Frame: Baseline (Day 0)
Measure: Count of Participants; unit: Participants
Arm/Group | Micropatch Application
Number analyzed (Participants) | 35
Participants
  L* ≤ 50 | 10
  L* 51-65 | 9
  L* > 65 | 16

4. Secondary Outcome: Hydration
Description: Baseline skin hydration will be measured using a capacitance probe. The software calculates arbitrary unitless values. Values less than 30 are considered very dry while values over 40 are considered sufficiently moisturized. Data are calculated as the mean of measurements from all 5 sites at each body location.
Time Frame: Baseline (Day 0)
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Micropatch Application
Number analyzed (Participants) | 35
unitless
  Forearm | 28.88 (8.3)
  Upper arm | 28.02 (8.94)
  Abdomen | 23.24 (8.5)

ADVERSE EVENTS:
Time Frame: Adverse Events were monitored at the micropatch sites during the 4 days while a subject was completing the study and for three days after study completion.
Description: Through the course of this study adverse events were recorded as reported from the subjects.
Arm/Group | Micropatch Application
All-Cause Mortality (participants affected / at risk) | 0/46
Serious Adverse Events (participants affected / at risk) | 0/46
Other Adverse Events (participants affected / at risk) | 3/46
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Micropatch Application (N=46)
Skin redness or irritation (Skin and subcutaneous tissue disorders) | 3 — Some skin redness or irritation was present where the medical tape had been in contact with the skin. All events resolved spontaneously after patch removal.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-24): https://cdn.clinicaltrials.gov/large-docs/77/NCT03657277/Prot_SAP_000.pdf